CLINICAL TRIAL: NCT07300007
Title: An Open-Label, Randomized, Crossover Study to Characterize the Pharmacokinetics and Relative Bioavailability of Liquid Metformin at 100 mg/mL and 250 mg/mL Compared With Standard Metformin Tablets
Brief Title: PK and Relative Bioavailability of Liquid Metformin vs Tablets in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ASP-016-MET
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: This is a single-arm, three-period, three-treatment crossover study in which all participants receive each metformin formulation in randomized sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Arm Crossover (Experimental)
  Interventions: Drug: Liquid Metformin 100 mg/mL; Drug: Liquid Metformin 250 mg/mL

INTERVENTIONS:
Drug: Liquid Metformin 100 mg/mL — A single oral dose of liquid metformin at a concentration of 100 mg/mL will be administered under fasting conditions in one treatment period of the crossover.
Drug: Liquid Metformin 250 mg/mL — A single oral dose of liquid metformin at a concentration of 250 mg/mL will be administered under fasting conditions in one treatment period of the crossover.

SUMMARY:
The study will evaluate the pharmacokinetics and relative bioavailability of two liquid metformin formulations (100 mg/mL and 250 mg/mL)

DETAILED DESCRIPTION:
The study will compare the pharmacokinetic profiles of two liquid metformin formulations (100 mg/mL and 250 mg/mL) with a standard metformin immediate-release tablet.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 to 55 years of age, inclusive.

Body mass index (BMI) between 18.0 and 30.0 kg/m², inclusive.

Medically healthy with no clinically significant findings on medical history, physical examination, vital signs, 12-lead ECG, or clinical laboratory tests, in the opinion of the investigator.

Non-smokers or light smokers (10 or fewer cigarettes per day or equivalent) willing to abstain from smoking during confinement.

Able to understand and provide written informed consent before any study procedures are conducted.

Willing and able to comply with all study requirements, including fasting restrictions and visit schedules.

Females of childbearing potential must use acceptable contraception as determined by the investigator.

Exclusion Criteria:

* Known hypersensitivity or contraindication to metformin or any excipients in the study formulations.

History or presence of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic, or psychiatric disorders that could affect study participation or data interpretation.

Estimated glomerular filtration rate (eGFR) less than 90 mL per minute per 1.73 square meters, or any clinically significant abnormal laboratory findings.

History of lactic acidosis.

Use of prescription medications, over-the-counter medications, herbal supplements, or dietary supplements within 14 days before first dosing, unless approved by the investigator.

Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV.

Positive urine drug test or positive alcohol breath test at screening or admission.

Participation in another clinical trial or receipt of an investigational product within 30 days or 5 half-lives (whichever is longer) before first study dose.

Blood donation of more than 450 mL or significant blood loss within 8 weeks before first dosing.

Pregnant or breastfeeding females.

Women of childbearing potential not using acceptable contraception.

Any condition that, in the opinion of the investigator, would make the participant unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to approximately 24 to 36 hours postdose in each treatment period
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC₀-t) | Up to approximately 24 to 36 hours postdose in each treatment period

IPD SHARING:
Plan to Share IPD: No